CLINICAL TRIAL: NCT01815034
Title: Transcutaneous Monitoring to Avoid Hypercapnea During Complex Catheter Ablations: a Joint Quality Initiative Pilot From Cardiac Electrophysiology and Anesthesiology
Brief Title: Trancutaneous Monitoring to Avoid Hypercapnea During Complex Catheter Ablations
Acronym: TCO2
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Dan Cantillon, Principal Investigator, The Cleveland Clinic
Other Study IDs: 13-083
Record Dates: First submitted 2013-03-12; First posted 2013-03-20 (Estimated); Last update posted 2014-08-19 (Estimated); Status verified 2013-03

CONDITIONS: Hypercapnia
MeSH Terms: conditions — Hypercapnia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Use of trancutaneous CO2 (TC02) monitoring to aide in titration of sedation of midazolam and fentanyl. Trancutaneous readings validated with invasively obtained specimens from existing arterial sheaths required during AF and VT ablations (trans-septal and retrograde aortic respectively)

DETAILED DESCRIPTION:
Cardiac electrophysiology procedures are typically performed under moderate (conscious) sedation in most centers. Advantages over general anesthesia include facilitating arrhythmia induction, avoidance of intubation and ventilator related complications and shorter post-procedure recovery times for most patients. However, the cumulative respiratory depressant effects of fentanyl and midazolam during prolonged procedures can rarely cause hypoventilation resulting in hypercapnea and respiratory failure. Complex catheter ablations for atrial fibrillation and ventricular tachycardia can exceed 3-5 hours in duration requiring large cumulative doses of midazolam and fentanyl. End tidal CO2 monitors, particularly in non-ventilated patients, have limitations and obtaining frequent arterial blood gas samples are often impractical. It remains unknown if contemporary trancutaneous CO2 monitoring (TCO2)can provide a feasible alternative to avoid over-sedation and resultant respiratory complications during complex catheter ablations with sufficient agreement to invasively obtained PCO2 data.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing catheter ablation for atrial fibrillation (AF) or ventricular tachycardia (VT) under moderate sedation.

Exclusion Criteria:

* Procedures scheduled for general anesthesia

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing catheter ablation for artial fibrillation or ventricular tachycardia
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2013-03; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Agreement with invasively obtained PCO2 data within 5 mm Hg | up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J Cantillon, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States